CLINICAL TRIAL: NCT04951999
Title: AssocIation of PULSatility and Occurrence of Complications Related to Mechanically Assisted Circulatory Support
Acronym: IMPULSMACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ICAN Nutrition Education and Research (Industry); University Hospital, Lille (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP190830; 2020-A01450-39 (Other: ANSM)
Record Dates: First submitted 2021-06-14; First posted 2021-07-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: End-stage Heart Failure
Keywords: LVAD; pulsatility index; Von Willebrand Factor
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Other)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — For 10 visits (out of the 12 of the protocol), ~40 ml of blood is sampled for research purposes in addition to care sampling.

SUMMARY:
The primary objective of this study is to determine whether preserved pulsatility for patients supported by CF-LVAD (continuous flow Left Ventricular Assist Device) is associated with less acquired deficiency of the Von Willebrand factor, a blood glycoprotein involved in hemostasis.

DETAILED DESCRIPTION:
Implantation of LVADs (Left Ventricular Assist Device) is a medium to long-term therapeutic option for patients with end-stage heart failure and isolated left ventricular dysfunction. Nevertheless, LVADs use remain limited by the frequency of their adverse effects, most of which being unpredictable. In the literature, loss of pulsatility seems to be associated with CF-LVADs complications, including bleeding. Accordingly, the primary objective of this study is to determine whether patient's preserved pulsatility is associated with less acquired deficiency of the Von Willebrand factor (VWF), a blood glycoprotein involved in hemostasis. This deficiency, characterized by a decrease or absence of VWF High Molecular Weight Multimers (HMWMs), is present to varying degrees in almost all patients with LVADs and is a major risk factor for bleeding complications in these patients. Pulsatility is estimated by the patient's blood pressure differential, measured 1) at discharge from the operating room (=transfer to care), 2) at discharge from care (=transfer to his or her room), 3) at discharge from the hospital (=transfer to rehabilitation), and then at each follow-up visit up to 6 months post-implantation. The primary endpoint is to determine whether a preserved pulsatility is associated with less acquired deficiency of the Von Willebrand factor ratio of High Molecular Weight Multimers (HMWMs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Patients for whom a decision to implant a left-sided monoventricular assist has been retained after discussion in the RCP of heart failure, transplantation and circulatory assistance (whatever the therapeutic strategy envisaged: waiting for transplantation, recovery or destination therapy).
3. Patients affiliated to a social security system (beneficiaries or beneficiaries entitled to benefits, excluding AME)
4. Signature of an informed consent by the patient or by the trusted person, or a close relative, if the patient is not able to do so

Exclusion Criteria:

1. Heart transplant patients
2. Patients who already had LVAD
3. Chronic renal failure patients on dialysis
4. Patients refusing to give informed consent
5. Patients deprived of liberty or under legal protection (guardianship, curators)
6. Pregnant or breastfeeding women
7. Ongoing participation in another intervention research protocol except LEVOECMO project (NCT04728932) and ANCHOR project (NCT04184635)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Von Willebrand factor high molecular weight multimers (HMWM) ratio | 30 days after LVAD IMPLANTATION
  Comparison of Von Willebrand factor high molecular weight multimers (HMWM) ratio at LVAD pre-implantation and at day 30.
  Measure of an correlation between preserved pulsatility and the HMWM ratio evolution during the first month after implantation.

SECONDARY OUTCOMES:
Severe postoperative gastrointestinal bleeding | 6 months
  Track record of patients undergoing gastrointestinal bleeding, identified by a decreased hemoglobin level associated with chronic iron deficiency anemia of unexplained cause and melena or bleeding demonstrated by exploration of the gastrointestinal tract by esophageal endoscopy, colonoscopy, or endoscopic videoscopy and resulting in any of the following:
  * Death
  * Re-operation
  * Hospitalization
  * An erythrocyte transfusion defined as:
    * Within 7 days of implantation :
  * Patients weighing 50 kg or more: ≥ 4U of packed red blood cells in a 24-hour period.
  * Patients weighing less than 50 kg: ≥ 20 mL/kg of packed red blood cells over a 24-hour period
    * After 7 days post-implantation : any transfusion of packed red blood cells.
Post-operative right ventricular failure | 6 months
  Track record of patients undergoing right ventricular failure, identified by:
  * Elevation of central venous pressure (CVP) >16 mmHg by direct or echocardiographic measurement (inferior vena cava diameter >20 mm and respiratory variations <50%) for more than 48 hours
  * and at least one of the following signs of hemodynamic failure persisting for more than 48 hours:
    * Increased inotropic score
    * Hyperlactatemia >3 mmol/l
    * Hepatic cytolysis: increase in AST and/or ALT by a factor of 3 or more after implantation
    * Degradation of renal function (AKIN grade 2: creatinine elevation > 50% compared with before explantation and diuresis < 0.5 ml/kg/24h for 12 hours)
    * Implantation of right temporary circulatory support (ECMO)
Platelet dysfunction | 6 months
  Platelet dysfunction defined by a significant increase in circulating levels of p-selectin and glycocalicin between pre- and post-implantation
Post-operative transient or permanent ischemic attack | 6 months
  Track record of patients undergoing ischemic attack (between 24 hours and 6 months post-operative) as assessed per INTERMACS definition
Vascular endothelium dysfunction | 6 months
  Vascular endothelial dysfunction defined by a significant increase in circulating levels of syndecan, thrombomodulin, TFPI and PAI-1 between pre- and post-implantation
Prolonged systemic inflammatory reaction syndrome | 6 months
  Monthly measures of following circulating inflammatory factors : TNFα et β, NF kappab, TGF α /β1/β2,IFNγ et β, IL-1β, IL-1RA, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p40, IL12-P70, IL-17, IL17A et F,CX3CL1 (fractalkine),MCP-1(CCL2), MIP-1 (CCL3), MIP-1β(CCL4), MIP-3-beta (CCL19), 6Ckine(CCL21), MCD (CCL22) Myostatin, calveolin-1.
Evolution of immune responses | 6 months
  Monthly phenotyping of monocytes and T cells
Aortic valve fusion | 6 months
  Monthly echographic evaluation
Aortic valve insufficiency | 6 months
  Monthly echographic evaluation
Evaluation of cardiac recovery | 6 months
  Monthly exercise stress test evaluation (starting 2 months post-operative)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEBRETON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupement Hospitalier pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.